CLINICAL TRIAL: NCT02698540
Title: A Prospective, Observational Study, of a High Calorie, Higher Protein Peptide Based Oral Nutrition Supplement (ONS) With Medium Chain Triglycerides (MCTs) in a Malnourished Population With GI Tolerance Impairment
Brief Title: A Study of an Oral Nutritional Supplement in a Malnourished Population With GI Tolerance Impairment
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA13
Record Dates: First submitted 2016-02-23; First posted 2016-03-03 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Nutritional Supplement — High calorie, high protein peptide based

SUMMARY:
The purpose is to observe the compliance to a high-calorie, high protein peptide-based nutritional supplement after 3 months in a malnourished population with impaired gastrointestinal tolerance living in nursing homes and as outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered malnourished, or is at risk for malnutrition based on MUST score ≥2.
* Subject is ≥18 years old.
* Subject has a condition that would benefit from a high calorie, higher protein ONS for GI tolerance impairment (e.g., diarrhea, nausea, vomiting, satiety or bloating).
* Subject conforms to the requirements set forth on the study product label.
* Subject is under the care of a health care professional for malnutrition and has recently (within the last 7 days prior to participating in this study) been prescribed 2 servings/day of the study ONS. Subject must have been naïve to ONS for GI tolerance impairment prior to being prescribed the study ONS.

Exclusion Criteria:

* The study physician determines the subject is not fit to participate
* Subject cannot provide informed consent to participate in the study.
* Subject cannot safely consume the oral nutritional supplement.
* Renal or liver failure (GFR< 60 ml/min or AST/ALTx3 normal) upper limit.
* Type 1 or type 2 diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include men and women who are free living (outpatient) or residing in a nursing home.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Study Product Compliance | Baseline to Week 12
  Subject reported diaries

SECONDARY OUTCOMES:
Body Weight | Baseline to Week 12
Nutrition Status | Baseline to Week 12
  Healthcare Professional completed screening
Quality of Life | Baseline to Week 12
  Subject reported questionnaire
Gastrointestinal Tolerance | Baseline to Week 12
  Subject reported scale
Body Mass Index | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sanz Barriuso, RD, PharmD, Study Chair — Abbott Nutrition
Locations (23):
- Spain (23):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital de Cruces 1758, Barakaldo
  - Hospital de Cruces 2029, Barakaldo
  - Hospital de Jerez, Cadiz
  - Hospital Universitario Reina Sofía de Córdoba, Córdoba
  - Hospital Universitario Campus de la Salud, Granada
  - Complejo Asistencial Universitario de Leon, Endocrinologia y Nutricion, León
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Principe de Asturias, Madrid
  - Hospital Universitario de Móstoles, Madrid
  - Hospital Costa del Sol 1740, Marbella
  - Hospital Costa del Sol 1743, Marbella
  - Centro Médico San Juan de la Cruz, Málaga
  - Hospital Rey Juan Carlos, Móstoles
  - Hospital General Universitario Reina Sofía de Murcia, Murcia
  - Hospital Vega Baja, Orihuela
  - Hospital del Bierzo, Ponferrada
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia 1695, Valencia
  - Hospital La Ribera, Valencia
  - Hospital de Vic, Vic
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No